CLINICAL TRIAL: NCT00322023
Title: PK/PD Study of Escalating Dose D-serine as Adjunctive Treatment in Schizophrenia
Brief Title: Safety and Effectiveness of D-serine in Schizophrenia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nathan Kline Institute for Psychiatric Research (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Daniel C. Javitt, MD, PhD, PI, National Institute of Mental Health (NIMH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: U01MH074356 (NIH); U01MH074356 (NIH); DATR A5-EPTD
Record Dates: First submitted 2006-05-02; First posted 2006-05-04 (Estimated); Results first posted 2020-10-05 (Actual); Last update posted 2020-10-05 (Actual); Status verified 2020-09

CONDITIONS: Schizophrenia
Keywords: Negative symptoms; NMDA; Glutamate; Glycine
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- D-serine 30 mg/kg (Experimental): D-serine 30 mg/kg
  Interventions: Drug: D-serine
- D-serine 60 mg/kg (Experimental): D-serine 60 mg/kg
  Interventions: Drug: D-serine
- D-serine 120 mg/kg (Experimental): D-serine 120 mg/kg
  Interventions: Drug: D-serine

INTERVENTIONS:
Drug: D-serine — D-serine at following dose levels: 30 mg/kg, 60 mg/kg, and 120 mg/kg. PK/PD studies done at day 1. Medication will be administered as powder dissolved in liquid given in two divided doses daily for 4 weeks.
Drug: D-serine
  Arms: D-serine 30 mg/kg
Drug: D-serine
  Arms: D-serine 60 mg/kg
Drug: D-serine
  Arms: D-serine 120 mg/kg

SUMMARY:
This study will determine whether increasing D-serine within the body will improve negative symptoms and cognitive impairments in people with schizophrenia.

DETAILED DESCRIPTION:
Schizophrenia is a life-long brain disorder affecting approximately 1 percent of Americans each year. Schizophrenia can be extremely disabling, causing people to hear voices, experience paranoia or hallucinations, believe that others are controlling their thoughts, and even fail at maintaining a job or caring for themselves. Current medications help to relieve most of these symptoms, but not all. Some people with schizophrenia still suffer from negative symptoms, such as difficulty with talking, expressing emotions, and motivation; they may also suffer from cognitive impairments, such as decreased concentration and memory loss. D-serine, an amino acid found within the body, activates brain cell receptors that appear to play a role in learning and memory. This study will determine whether adding a D-serine solution to a stable antipsychotic medication regimen will decrease negative symptoms in people with schizophrenia.

Participants in this open-label study will remain on their regular medication regimen for at least 2 weeks. During this time and before starting treatment, participants will be interviewed about their emotional problems, marital status, education, family background, employment history, and any drug or alcohol problems. Participants will also undergo a physical exam, an electrocardiogram (EKG), vital sign measurements, psychological tests, cognitive tasks, and an electroencephalogram (EEG). Participants will then begin 4 weeks of treatment with D-serine. In addition to participants' regular medication regimen, they will drink a D-serine powder mixed with water twice daily. Every 2 weeks, participants will undergo a physical exam and an interview about any changes in symptoms or emotional problems that they may be experiencing. Blood and urine samples will be taken throughout the study. After 4 weeks, participants will undergo an EKG, EEG, and the same psychological tests and cognitive tasks completed prior to treatment. A follow-up visit will occur 2 weeks post-treatment to monitor any changes in negative symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Structured Clinical Interview for DSM-III-R diagnosis of schizophrenia or schizoaffective disorder
* PANSS 3 factor negative symptom inclusion score greater than 20 prior to study entry
* PANSS total score between 60 and 110
* Simpson-Angus Scale total score of 12 or less
* Calgary Depression Inventory total score of 10 and suicide score less than 2
* No change in Clinical Global Impressions (CGI) Scale score prior to study entry
* Chlorpromazine (CPZ) equivalent of 1500 or less
* Willing to use an effective form of birth control throughout the study if sexually active

Exclusion Criteria:

* High extrapyramidal symptom (EPS) levels
* Began, discontinued, or adjusted psychotropic medication within 2 weeks of study entry
* Taking investigational medication within 2 weeks of study entry
* Contraindication to study medication
* Serious or unstable medical illness
* Pregnant or breastfeeding
* Alcohol or drug abuse within 6 months of study entry
* Diagnosed with neurodegenerative disease or a seizure disorder
* History of a kidney impairment
* Currently taking clozapine
* Currently taking more than two antipsychotic medications
* Currently taking stimulants or cholinesterase inhibitors

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 55 (Actual)
Dates: Start 2006-03; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel C. Javitt, MD, PhD, Principal Investigator — Nathan Kline Institute
Locations (3):
- United States (3):
  - Yale University School of Medicine, New Haven, Connecticut
  - The Zucker Hillside Hospital, Glen Oaks, New York
  - The Nathan S. Kline Institute for Psychiatric Research, Orangeburg, New York

REFERENCES:
- [Derived] Kantrowitz JT, Epstein ML, Lee M, Lehrfeld N, Nolan KA, Shope C, Petkova E, Silipo G, Javitt DC. Improvement in mismatch negativity generation during d-serine treatment in schizophrenia: Correlation with symptoms. Schizophr Res. 2018 Jan;191:70-79. doi: 10.1016/j.schres.2017.02.027. Epub 2017 Mar 18. PMID 28318835

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Nathan Kline Institute, Yale University, Zucker Hillside
Groups:
- D-serine 30 mg/kg; D-serine 60 mg/kg; D Serine 120 mg/kg: Open label, adjunctive to antipsychotics for 4 weeks
Period: Overall Study
Arm/Group | D-serine 30 mg/kg | D-serine 60 mg/kg | D Serine 120 mg/kg
Started | 12 | 21 | 22
Completed | 12 | 19 | 16
Not Completed | 0 | 2 | 6
Not completed — various | 0 | 2 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | D-serine 30 mg/kg | D-serine 60 mg/kg | D Serine 120 mg/kg | Total
Number analyzed (Participants) | 12 | 21 | 22 | 55
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 12 | 21 | 22 | 55
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.7 (11.4) | 43.9 (9.4) | 43.2 (9.6) | 43 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 4 | 11
  Male | 9 | 17 | 18 | 44

OUTCOME MEASURES:

1. Primary Outcome: Renal Safety Measures
Description: number of renal adverse events (serum and urinalysis)
Time Frame: Measured at Week 4
Population: study completers
Measure: Number; unit: adverse events
Groups:
- D-serine 30 mg/kg; D-serine 60 mg/kg; D Serine 120 mg/kg: 4 weeks of adjunctive treatment
Arm/Group | D-serine 30 mg/kg | D-serine 60 mg/kg | D Serine 120 mg/kg
Number analyzed (Participants) | 12 | 19 | 16
adverse events | 0 | 0 | 1

2. Secondary Outcome: Positive and Negative Symptoms Scale (PANSS)
Description: Absolute Change in PANSS over four weeks (change between baseline and final measurements). The PANSS is a 30-item rating scale widely used in assessment of medication effects in schizophrenia. The PANSS ranges from 30-210, with lower scores showing less symptoms. Larger change is better.
Time Frame: Measured at Week 4
Population: Study completers
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | D-serine 30 mg/kg | D-serine 60 mg/kg | D Serine 120 mg/kg
Number analyzed (Participants) | 12 | 19 | 16
units on a scale | 5.1 (5.3) | 4.4 (8.9) | 6.3 (5.5)
Statistical Analysis 1: Comparison: D-serine 30 mg/kg; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; These are paired t test baseline vs final for the 30 mg/kg dose
Statistical Analysis 2: Comparison: D-serine 60 mg/kg; Test type: Superiority; p < 0.05, t-test, 2 sided; These are paired t test baseline vs final for the 60 mg/kg dose
Statistical Analysis 3: Comparison: D Serine 120 mg/kg; Test type: Superiority — These are paired t test baseline vs final for the 120 mg/kg dose; p < 0.01, t-test, 2 sided

3. Secondary Outcome: Measurement and Treatment Research to Improve Cognition in Schizophrenia (MATRICS) Battery
Description: Change over 4 weeks. The MATRICS is a scale measuring cognition, and reported as T-score, with 50 as the population average and every 10 points representing a change of 1 standard deviation from the population average. Higher scores represent an improvement
Time Frame: Measured at Week 4
Population: study completers
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | D-serine 30 mg/kg | D-serine 60 mg/kg | D Serine 120 mg/kg
Number analyzed (Participants) | 12 | 19 | 16
units on a scale | 0.8 (3.0) | 3.9 (3.5) | 2.8 (2.8)
Statistical Analysis 1: Comparison: D-serine 30 mg/kg; Test type: Superiority or Other; p = 0.39, t-test, 2 sided — These are paired t test baseline vs final for 30mg/kg
Statistical Analysis 2: Comparison: D-serine 60 mg/kg; Test type: Superiority; p < 0.001, t-test, 2 sided — These are paired t test baseline vs final for 60mg/kg
Statistical Analysis 3: Comparison: D Serine 120 mg/kg; Test type: Superiority; p = 0.01, t-test, 2 sided — These are paired t test baseline vs final for 120mg/kg

ADVERSE EVENTS:
Arm/Group | D-serine 30 mg/kg | D-serine 60 mg/kg | D Serine 120 mg/kg
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/19 | 1/16
Other Adverse Events (participants affected / at risk) | 0/12 | 0/19 | 2/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | D-serine 30 mg/kg (N=12) | D-serine 60 mg/kg (N=19) | D Serine 120 mg/kg (N=16)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) — 2+ proteinuria without glycosuria during the final week of treatment with no significant change in creatinine that resolved following dserine discontinuation.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | D-serine 30 mg/kg (N=12) | D-serine 60 mg/kg (N=19) | D Serine 120 mg/kg (N=16)
asymptomatic transaminitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 2 (2)

LIMITATIONS AND CAVEATS:
Open Label

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No